CLINICAL TRIAL: NCT03387410
Title: Safety and Efficacy of IRDye 800BK in Ureter Identification Via Fluorescence Detection During Laparoscopic Abdominal Surgery
Brief Title: Ureter Identification With IRDye 800BK
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Oxford University Hospitals NHS Trust (Other)
Collaborators: University of Oxford (Other)
Responsible Party: Principal Investigator, Thomas Barnes, Clinical Research Fellow, Oxford University Hospitals NHS Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 12932
Record Dates: First submitted 2017-12-18; First posted 2018-01-02 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Ureter Injury
Keywords: Laparoscopic surgery; Fluorescence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intravenous IRDye 800BK (Experimental): Patients undergoing laparoscopic bowel resection & laparoscopic donor nephrectomy
  Interventions: Drug: Intravenous IRDye 800BK

INTERVENTIONS:
Drug: Intravenous IRDye 800BK — Fluorescence of the ureter using IRDye 800BK

SUMMARY:
Phase 1/2a study, second in-man utilising IRDye800BK in ureteric identification using fluorescence throughout abdominal surgery. Study is open label, non-randomised prospective study.

ELIGIBILITY:
Inclusion Criteria (Group A & B participants)

* Participant is willing and able to give informed consent for participation in the trial.
* Male or Female, aged 18 years or above.
* Undergoing elective laparoscopic abdominal surgery or undergoing planned laparoscopic donor nephrectomy (donation)
* Participant has available laboratory and ECG results within 3 months of enrolment.
* Female participants of child bearing potential and male participants whose partner is of child bearing potential must be willing to ensure that they or their partner use effective contraception during the trial and for 3 months thereafter
* In the Investigator's opinion, is able and willing to comply with all trial requirements.
* Group A only: Participant is undergoing laparoscopic colorectal surgery
* Group B only: Participant is undergoing laparoscopic donor nephrectomy

Exclusion Criteria (Group A & B participants)

The participant may not enter the trial if ANY of the following apply:

* Female participant who is pregnant, lactating or planning pregnancy throughout the trial.
* Significant renal impairment (eGFR of under 50mL/min/1,73m2)
* Significant liver impairment as defined as:

  * AST > 3.0 x ULN or
  * ALT > 3.0 x ULN or
  * Total serum bilirubin > 1.5 x ULN
* Participants involved with another research trial involving an unlicensed medicine in the past 12 weeks.
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.
* Known allergy to D-Mannitol or citric acid
* Group B Only: Laparoscopic donor nephrectomy patients in whom the kidney recipient has refused participation or if the recipient is being transplanted in another transplant centre

Inclusion criteria for transplant recipients

* Participant must be willing and able to give informed consent for trial participation
* Male or female aged 18 years or over
* Is able and willing to comply with all trial requirements
* Receiving a kidney from a participant recruited to this study

Exclusion criteria for transplant recipients

• Female who is pregnant, lactating, or planning pregnancy throughout the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-04-06 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-16 (Actual)

PRIMARY OUTCOMES:
Change of signal to background measurements and visualisation of fluorescence in the ureter | 0, 5, 10, 20, 30, 40, 50, 60, 70, 80, 90, 100, 120, 180, 240 minutes post dose
  Signal to background is an objective measurement of fluorescence signal
Change in subjective assessment of ureter visualisation with and without fluorescence | 0, 5, 10, 20, 30, 40, 50, 60, 70, 80, 90, 100, 120, 180, 240 minutes post dose

SECONDARY OUTCOMES:
Number of adverse events related to IRDye 800BK administration | 30 days post administration

CONTACTS AND LOCATIONS:
Locations (1):
- Oxford University Hospitals NHS Foundation Trust, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No